CLINICAL TRIAL: NCT05898529
Title: Prevalence of Asymptomatic COVID-19 Infection in Pediatric Surgical Patients
Brief Title: COVID Infection in Pediatric Surgical Patient
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAnes2023 Paed COVID Afr
Record Dates: First submitted 2023-06-09; First posted 2023-06-12 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid antigen test — COVID-19 rapid antigen testing of nasal swab

SUMMARY:
Children infected with COVID-19 are mostly asymptomatic. There is a dearth of data on the epidemiology of COVID-19 in the pediatric population. This is a prospective observational clinical study of pediatric surgical patients. COVID-19 rapid antigen testing will be performed on pediatric patients.

DETAILED DESCRIPTION:
Children infected with COVID-19 are mostly asymptomatic or mildly symptomatic. Children may spread COVID-19 to the elderly, vulnerable patients and medical staff. There is a dearth of data on the epidemiology of COVID-19 in the pediatric surgical population. Rapid antigen detection tests for the diagnosis of COVID-19 are reliable, simple, fast, and inexpensive.

This is a prospective observational clinical study. The study population will include all consenting pediatric surgical patients, aged 2-17 years. Informed consent will be obtained from each patient and the legal guardian who agree to participate in the study. Nasopharyngeal swab specimens will be collected from anesthetized pediatric patients. COVID-19 rapid antigen testing will be performed according to the equipment manufacturer's instructions.

Data collection will include COVID-19 test result, nasal swab complication, patient demographics, surgical history, medical history, regular medications, COVID-19 symptoms, and COVID-19 exposure information. COVID-19 symptoms that will be recorded are cough, wheeze, nasal congestion, breathing difficulty, new loss of taste or smell, fever, chills, rigors, body aches, sore throat, nausea, and fatigue. COVID-19 exposure will be considered as being within 6 feet of a person with diagnosed COVID-19 infection in the previous 14 days.

ELIGIBILITY:
Inclusion Criteria:

* surgical patients aged 2-17 years
* informed consent for surgery
* no COVID-19 diagnosis in previous 6 months
* no history of nasal bleeding
* no history of coagulopathy.

Exclusion Criteria:

* patient refusal of testing
* difficulty in obtaining consent
* COVID-19 diagnosis in recent 6 month
* history of nasal bleeding
* history of coagulopathy.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Consecutive surgical patients, aged 2-17 years.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Antigen test positive result | 1 day
  COVID-19 antigen test positive

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No